CLINICAL TRIAL: NCT03346759
Title: Examining the Impact of Tampon Use on the Vaginal Microbiota
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jason Bell, MD, MPH, MS, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00122922
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Results first posted 2018-07-20 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: Vaginal Microbiota
Keywords: tampon; menstruation; menstrual period

STUDY DESIGN:
Intervention Model Description: Subjects were provided with 24 Tampax Pearl Regular Tampons (tampon A) to use exclusively for one of the first two menstrual cycles during the study. Subjects were provided with 24 Playtex Gentle Glide 360 Regular Tampons (tampon B) to use exclusively for the other of the first two menstrual cycle during the study. Subjects used tampons A and B in a randomly assigned order. Subjects then used tampons of their choosing for the third menstrual cycle of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tampon A First (Experimental): Subjects were provided with 24 Tampax Pearl Regular Tampons (tampon A) to use exclusively for the first of two consecutive menstrual cycles. Subjects were then provided with 24 Playtex Gentle Glide 360 Regular Tampons (tampon B) to use exclusively for the second of two consecutive menstrual cycles. For the third menstrual cycle, subject used tampons of their choosing.
  Interventions: Device: Tampon A; Device: Tampon B
- Tampon B First (Experimental): Subjects were provided with 24 Playtex Gentle Glide 360 Regular Tampons (tampon B) to use exclusively for the first of two consecutive menstrual cycles. Subjects were then provided with 24 Tampax Pearl Regular Tampons (tampon A) to use exclusively for the second of two consecutive menstrual cycles. For the third menstrual cycle, subject used tampons of their choosing.
  Interventions: Device: Tampon A; Device: Tampon B

INTERVENTIONS:
Device: Tampon A — 24 Tampax Pearl Regular Tampons for use during a single menstrual period.
Device: Tampon B — 24 Playtex Gentle Glide 360 Regular Tampons for use during a single menstrual period.

SUMMARY:
The vaginal microbiota is the community of bacteria in the vagina. The composition of the vaginal microbiota (which bacteria are present and how many of each are present) is known to affect vaginal health and contribute to the development of bacterial vaginosis (the largest cause of vaginal discharge and malodor, and the most common vaginal disorder). It is also known that the composition of the vaginal microbiota changes across a menstrual cycle with the largest changes happening during a woman's period. However, it is not know how tampon use affects vaginal microbiota composition. This study is being done to learn what effect tampon use has on vaginal microbiota composition during a woman's period and between periods.

ELIGIBILITY:
Inclusion Criteria:

* regular menstrual cycles lasting 21-35 days
* menses lasting for at least 4 days
* current tampon user
* good self-reported general health
* good self-reported vaginal health

Exclusion Criteria:

* currently pregnant
* planning to become pregnant in 4 months following enrollment
* difficulty using tampons
* current toxic shock syndrome
* history of toxic shock syndrome
* current sexually transmitted infection
* current urinary tract infection
* currently using antibiotics
* antibiotic use in 4 weeks prior to enrollment
* current antifungal use
* antifungal use in 4 weeks prior to enrollment
* autoimmune condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2017-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Bell, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Enrollment to Baseline Data Collected
Arm/Group | Tampon A First | Tampon B First
Started | 15 | 13
Completed | 13 (Participants assigned to the Tampon A First arm who provided at least one vaginal microbiota sample.) | 10 (Participants assigned to the Tampon B First arm who provided at least one vaginal microbiota sample.)
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3
Period: First Menstrual Cycle
Arm/Group | Tampon A First | Tampon B First
Started | 13 | 10
Completed | 12 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Menstrual Cycle
Arm/Group | Tampon A First | Tampon B First
Started | 12 | 10
Completed | 11 | 10
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Third Menstrual Cycle
Arm/Group | Tampon A First | Tampon B First
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who provided at least one vaginal microbiota sample.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tampon A First | Tampon B First | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (5.0) | 24.3 (4.0) | 26.1 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic white | 10 | 8 | 18
  Asian | 1 | 0 | 1
  Hispanic | 0 | 2 | 2
  Black | 0 | 0 | 0
  Other | 2 | 0 | 2
Relative abundance of Lactobacillus species [Median (Inter-Quartile Range); unit: relative abundance] — Relative abundance is defined as the proportion of total identified bacteria in a sample that are a given type of bacteria. The Lactobacillus species included here are L. crispatus, L. iners, L. gasseri, and L. jensenii. Thus, a relative abundance of Lactobacillus species equal to 0.9 would mean that 90% of the bacteria identified in a sample are Lactobacillus species.
  relative abundance | .9667 [.9192 to .9898] | .9727 [.9521 to .9877] | .9705 [.9301 to .9894]
Relative abundance of Gardnerella vaginalis [Median (Inter-Quartile Range); unit: relative abundance] — Relative abundance is defined as the proportion of total identified bacteria in a sample that are a given type of bacteria. Thus, a relative abundance of Gardnerella vaginalis equal to 0.9 would mean that 90% of the bacteria identified in a sample are Gardnerella vaginalis.
  relative abundance | .000091 [0 to .000094] | .000019 [0 to .000136] | .000045 [0 to .000499]

OUTCOME MEASURES:

1. Primary Outcome: Change in Relative Abundance of Lactobacillus Species
Description: The differences in relative abundance of Lactobacillus species between: the last swab collected during menstrual cycle 1 and the first swab collected, the last swab collected during menstrual cycle 2 and the first swab collected, and the last swab collected during menstrual cycle 3 and the first swab collected. Relative abundance is defined as the proportion of total identified bacteria in a sample that are a given type of bacteria. The Lactobacillus species included here are L. crispatus, L. iners, L. gasseri, and L. jensenii. Thus, a relative abundance of Lactobacillus species equal to 0.9 would mean that 90% of the bacteria identified in a sample are Lactobacillus species.
Time Frame: Baseline, end of first menstrual cycle (approximately 6 weeks), end of second menstrual cycle (approximately 10 weeks), and end of third menstrual cycle (approximately 14 weeks)
Population: Participants analyzed are those that provided samples through the end of the given menstrual cycle.
Measure: Median (Inter-Quartile Range); unit: relative abundance
Arm/Group | Tampon A First | Tampon B First
Number analyzed (Participants) | 12 | 10
relative abundance
  Baseline to end of first cycle | .0084 [-.0017 to .0274] | -.0014 [-.0148 to .0242]
  Baseline to end of second cycle: number analyzed (Participants) | 11 | 10
  Baseline to end of second cycle | -.00004 [-.0121 to .0368] | .0104 [-.0346 to .0354]
  Baseline to end of third menstrual cycle: number analyzed (Participants) | 11 | 10
  Baseline to end of third menstrual cycle | -.0350 [-.1723 to .0304] | .0238 [.0107 to .0349]

2. Secondary Outcome: Change in Relative Abundance of Gardnerella Vaginalis
Description: The differences in relative abundance of Gardnerella vaginalis between: the last swab collected during menstrual cycle 1 and the first swab collected, the last swab collected during menstrual cycle 2 and the first swab collected, and the last swab collected during menstrual cycle 3 and the first swab collected. Relative abundance is defined as the proportion of total identified bacteria in a sample that are a given type of bacteria. Thus, a relative abundance of Gardnerella vaginalis equal to 0.9 would mean that 90% of the bacteria identified in a sample are Gardnerella vaginalis.
Time Frame: as for outcome 1
Population: Participants analyzed are those that provided samples through the end of the given menstrual cycle.
Measure: Median (Inter-Quartile Range); unit: relative abundance
Arm/Group | Tampon A First | Tampon B First
Number analyzed (Participants) | 12 | 10
relative abundance
  Baseline to end of first cycle | .000046 [-.000303 to .004230] | 0 [-.000124 to 0]
  Baseline to end of second cycle: number analyzed (Participants) | 11 | 10
  Baseline to end of second cycle | -.000045 [-.000788 to .001620] | 0 [-.000115 to 0]
  Baseline to 14 weeks: number analyzed (Participants) | 11 | 10
  Baseline to 14 weeks | -.000045 [-.004297 to .000030] | 0 [-.000124 to .000075]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of study participation for each subject (baseline window and menstrual cycles 1, 2, and 3; approximately 14 weeks per subject).
Groups:
- Tampon A: All participants while using Tampax Pearl Regular Tampons regardless of tampon sequence.
- Tampon B: All participants while using Playtex Gentle Glide 360 Regular Tampons regardless of tampon sequence.
- Tampon of Choice (Third Period): All participants during the third menstrual cycle.
Arm/Group | Tampon A | Tampon B | Tampon of Choice (Third Period)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT03346759/Prot_SAP_000.pdf